CLINICAL TRIAL: NCT04003675
Title: Sexual Harassment Among Students at Elite Sport High Schools and Regular High Schools in Norway
Brief Title: Sexual Harassment Within and Outside Sports
Status: Completed | Type: Observational
Sponsor: Norwegian School of Sport Sciences (Other)
Collaborators: The Norwegian Women´s Public Health Association (Other); Norwegian Extra Foundation for Health and Rehabilitation (Other); University of Agder (Other); University of Toronto (Other); UiT The Arctic University of Norway (Other)
Responsible Party: Principal Investigator, Professor Jorunn Sundgot-Borgen, Professor, Norwegian School of Sport Sciences
Other Study IDs: 2019/FO244849
Record Dates: First submitted 2019-06-27; First posted 2019-07-01 (Actual); Last update posted 2021-11-03 (Actual); Status verified 2021-11

CONDITIONS: Sexual Harassment; Sexual Abuse; Psychological Distress; Prevention
MeSH Terms: conditions — Sexual Harassment

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Adolescent elite athletes: Adolescent boys and girls elite athletes over 16 years of age studying at elite sport high schools in Norway.
- Adolescent controls: Adolescent boys and girls over 16 years of age studying at regular high schools in Norway.
- Trainers and leaders: Trainers (with more than 20 percent employment status) at elite sport high schools, and leaders/principals at elite sport high schools and regular high schools.

SUMMARY:
This study examines sexual harassment and abuse in and outside sports among adolescent elite athlete boys and girls, adolescent control students, trainers and leaders at elite sport high schools and regular high schools in Norway.

DETAILED DESCRIPTION:
The purpose of the study is to examine the prevalence and outcome of sexual harassment within and outside sports, including who the perpetrators are, the association between experienced sexual harassment and psychological health, knowledge of report mechanisms and emergency plans, and the participants suggestions for preventive strategies. The knowledge from this study will be a good basis to establish and implement prevention strategies and educational programs in the future.

Students, trainers (with more than 20 % employment status) and leaders at elite sport high schools and regular high schools in Norway will answer a questionnaire at two measurement points. Additionally, a sample of randomly selected students who report experiences with sexual harassment, and a random sample of trainers and leaders, will be invited to participate in an individual in-depth interview. Students scoring above cut-off on the questionnaire measuring symptoms of eating disorders (EDE-q) will be invited to a separate diagnostic interview (EDE).

A group of students will also participate in a test-retest examination of the reliability of the questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Over 16 years of age
* Students in 2nd grade elite sport high schools in Norway
* Students in 2nd grade at regular high schools (no specialization) in Viken and Oslo in Norway
* Trainers with more than 20 percent employment status at elite sport highs schools
* Leaders/principles at the attending elite sport- and regular high schools

Exclusion Criteria:

* Students under 16 years of age
* Trainers with less than 20 percent employment status
* Students/trainers not understanding written Norwegian language

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Students:
  Students in 2nd grade at public and private elite sport high schools in Norway, and a corresponding number of reference students in 2nd grade at representative regular high schools (no sport specialization) in the counties Viken and Oslo in Norway.
  Trainers and leaders:
  All administrative responsible employees (principles/inspectors) at public and private elite sport high schools and regular high schools, in addition to trainers at elite sport high schools with more than 20 % employment status.
Sampling Method: Non-Probability Sample
Enrollment: 1250 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2021-10-12 (Actual); Study Completion 2021-10-12 (Actual)

PRIMARY OUTCOMES:
Sexual harassment | Baseline
  Adolescent elite athletes and controls will answer a self-reported questionnaire regarding prevalence of sexual harassment, awareness of reporting mechanisms and emergency plans, suggestions for how to prevent sexual harassment.
Sexual harassment | 1 year after baseline
  Adolescent elite athletes and controls will answer a self-reported questionnaire regarding prevalence of sexual harassment, awareness of reporting mechanisms and emergency plans, suggestions for how to prevent sexual harassment.
Sexual harassment | Two weeks (test-retest)
  Adolescent elite athletes and controls will answer a self-reported questionnaire regarding prevalence of sexual harassment, awareness of reporting mechanisms and emergency plans, suggestions for how to prevent sexual harassment.

SECONDARY OUTCOMES:
Symptoms of eating disorders | Baseline
  Adolescent elite athletes and controls will answer the self-reported questionnaire "Eating Disorder Examination Questionnaire-6". The questionnaire consists of 28 items measuring symptoms and severity of eating disorders.
Symptoms of eating disorders | 1 year after baseline
  Adolescent elite athletes and controls will answer the self-reported questionnaire "Eating Disorder Examination Questionnaire-6". The questionnaire consists of 28 items measuring symptoms and severity of eating disorders.
Symptoms of eating disorders | Two weeks (test-retest)
  Adolescent elite athletes and controls will answer the self-reported questionnaire "Eating Disorder Examination Questionnaire-6". The questionnaire consists of 28 items measuring symptoms and severity of eating disorders.
Health related quality of life | Baseline
  Adolescent elite athletes and controls will answer two questions from the self-reported questionnaire "The World Health Organization Quality of Life Assessment Instrument" (WHOQOL-BREF). The items measure overall perception of quality of life and overall satisfaction with own health during the last two weeks on a 5-point Likert-scale ranging from very poor/very dissatisfied to very good/very satisfied.
Health related quality of life | 1 year after baseline
  Adolescent elite athletes and controls will answer two questions from the self-reported questionnaire "The World Health Organization Quality of Life Assessment Instrument" (WHOQOL-BREF). The items measure overall perception of quality of life and overall satisfaction with own health during the last two weeks on a 5-point Likert-scale ranging from very poor/very dissatisfied to very good/very satisfied.
Health related quality of life | Two weeks (test-retest)
  Adolescent elite athletes and controls will answer two questions from the self-reported questionnaire "The World Health Organization Quality of Life Assessment Instrument" (WHOQOL-BREF). The items measure overall perception of quality of life and overall satisfaction with own health during the last two weeks on a 5-point Likert-scale ranging from very poor/very dissatisfied to very good/very satisfied.
Resilience | Baseline
  Adolescent elite athletes and controls will answer the self-reported questionnaire "The Resilience Scale for Adolescents (READ)" measuring their ability to handle stress and negative life events. The participants are asked to indicate how much they agree or disagree to 28 items using a 5-point Likert scale.
Resilience | 1 year after baseline
  Adolescent elite athletes and controls will answer the self-reported questionnaire "The Resilience Scale for Adolescents (READ)" measuring their ability to handle stress and negative life events. The participants are asked to indicate how much they agree or disagree to 28 items using a 5-point Likert scale.
Resilience | Two weeks (test-retest)
  Adolescent elite athletes and controls will answer the self-reported questionnaire "The Resilience Scale for Adolescents (READ)" measuring their ability to handle stress and negative life events. The participants are asked to indicate how much they agree or disagree to 28 items using a 5-point Likert scale.
Self-esteem | Baseline
  Adolescent elite athletes and controls will answer the self-reported questionnaire "Rosenberg self-esteem scale" (RSES) consisting of 10 items measuring global self-esteem related to overall feelings of self-worth and self-acceptance. The participants are asked to indicate how much they agree or disagree to the items using a 4-point Likert scale ranging from strongly agree to strongly disagree.
Self-esteem | 1 year after baseline
  Adolescent elite athletes and controls will answer the self-reported questionnaire "Rosenberg self-esteem scale" (RSES) consisting of 10 items measuring global self-esteem related to overall feelings of self-worth and self-acceptance. The participants are asked to indicate how much they agree or disagree to the items using a 4-point Likert scale ranging from strongly agree to strongly disagree.
Self-esteem | Two weeks (test-retest)
  Adolescent elite athletes and controls will answer the self-reported questionnaire "Rosenberg self-esteem scale" (RSES) consisting of 10 items measuring global self-esteem related to overall feelings of self-worth and self-acceptance. The participants are asked to indicate how much they agree or disagree to the items using a 4-point Likert scale ranging from strongly agree to strongly disagree.
Subjective health complaints | Baseline
  Adolescent elite athletes and controls will answer the self-reported questionnaire "Health Behavior in School Children" measuring how often they have experienced 8 different physical and psychological health complaints (on a five-point scale ranging from almost every day to seldom/never) during the last 6 months.
Subjective health complaints | 1 year after baseline
  Adolescent elite athletes and controls will answer the self-reported questionnaire "Health Behavior in School Children" measuring how often they have experienced 8 different physical and psychological health complaints (on a five-point scale ranging from almost every day to seldom/never) during the last 6 months.
Subjective health complaints | Two weeks (test-retest)
  Adolescent elite athletes and controls will answer the self-reported questionnaire "Health Behavior in School Children" measuring how often they have experienced 8 different physical and psychological health complaints (on a five-point scale ranging from almost every day to seldom/never) during the last 6 months.
Sexual harassment experiences from trainers | Baseline
  Trainers and leaders will answer a questionnaire regarding their experiences with incidents of sexual harassment, awareness of reporting mechanisms and emergency plans, suggestions for how to prevent sexual harassment.
Sexual harassment interview | Baseline
  In-depth interviews with students, trainers and leaders about their experiences with sexual harassment, awareness of reporting mechanisms and suggestions for how to prevent sexual harassment in the future.
Eating disorder examination (EDE) interview | Following the 1 year-follow up questionnaire
  Students scoring above cut-off on the questionnaire EDE-q at the 1-year follow up questionnaire will be invited to a diagnostic interview (EDE) measuring eating disorder psychopathology/diagnosis.

CONTACTS AND LOCATIONS:
Overall Officials: Jorunn Sundgot-Borgen, PhD, Study Chair — Norwegian School of Sport Sciences
Locations (1):
- Norwegian school of sport sciences, Oslo, Norway

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Sundgot-Borgen C, Sundgot-Borgen J, Solvberg N, Torstveit MK, Mountjoy M, Mathisen TF. Factors predicting disordered eating and the prevalence of eating disorders in adolescent elite athletes, trained athletes and a reference group: a prospective controlled two-step study. Br J Sports Med. 2025 Jul 17;59(15):1043-1054. doi: 10.1136/bjsports-2024-108808. PMID 40097165